CLINICAL TRIAL: NCT05463393
Title: Humulus Lupus Extract Rich in Xanthohumol Improves Clinical Course in Critically Ill COVID-19 Patients
Brief Title: Xanthohumol as an Adjuvant Therapy in Critically Ill COVID-19 Patients
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: We are waiting for the additional founds.
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Wojciech Dąbrowski, Prof MD PhD, Head of Chair and First Department of Anaesthesiology and Intensive Therapy, Medical University of Lublin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DS352/2020
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-12

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Intervention Model Description: Patients were randomized in a double-blind, placebo-controlled fashion into two groups using sealed envelopes
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Xn (Experimental): Patients who received extract from Humulus lupus L rich in Xanthohumol (Hop-RXn™, BioActive-Tech Ltd, Lublin, Poland; http://xanthohumol.com.pl/) as an adjuvant therapy. Based on pharmacokinetics and bioactivity, Xn was administered enterally three times a day every 8 hours at a dose of 1.5 mg/kg body weight (4.5 mg/kg body weight/day) for 7 days. The first dose of Xn was administered within 4 hours after admission to the ICU.
  Interventions: Biological: Xanthohumol - prenylated chalcone extracted from female inflorescences of hop cones (Humulus lupus). Hop-RXn™, BioActive-Tech Ltd, Lublin, Poland; http://xanthohumol.com.pl/
- Group C (Placebo Comparator): Patients who received 0.9% NaCl at the oral volume 1 mL (similar to Xn volume) three times a day every 8 hours. The first dose of Xn was administered within 4 hours after admission to the ICU.
  Interventions: Biological: Xanthohumol - prenylated chalcone extracted from female inflorescences of hop cones (Humulus lupus). Hop-RXn™, BioActive-Tech Ltd, Lublin, Poland; http://xanthohumol.com.pl/

INTERVENTIONS:
Biological: Xanthohumol - prenylated chalcone extracted from female inflorescences of hop cones (Humulus lupus). Hop-RXn™, BioActive-Tech Ltd, Lublin, Poland; http://xanthohumol.com.pl/ — The appropriate dose of Xanthohumol was solved in 1 mL of propylene glycol

SUMMARY:
It has been well documented that coronavirus COVID-19 disease is associated with massive inflammatory response and cytokine storm. Several medications have been used to ameliorate COVID-19-related inflammation. Xanthohumol, a natural medication extracted from hop cones, possesses strong anti-inflammatory properties and can reduce the severity of inflammatory response. The aim of this study is to analyze the effect of Xanthohumol on clinical course, inflammatory response and outcome in patients admitted to the ICU due to COVID-related acute respiratory failure with an oxygenation index (PaO2/FiO2) less than 150.

DETAILED DESCRIPTION:
Xanthohumol inhibits proinflammatory pathways in different independent mechanisms. Ir inhibits farnesoid X receptor activity, and reduces the synthesis and release of different proinflammatory cytokines such as IL-1β, IL-6, IL-8, IL-12p70, TNFα and interferon γ. The pathomechanism of its anti-inflammatory activity is associated with the suppression of nuclear factor-kappa B. Additionally, Xanthohumol inhibits inflammatory-induced endothelial disorders, which are associated with an improvement in blood velocity and a reduction in the risk of arterial thrombosis, especially in pulmonary arteries. An increase in proinflammatory release, known as cytokine storm, as well as increased incidences of vascular thrombosis, are observed in coronavirus infection. Hence, Xanthohumol may reduce the severity of the clinical course in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of COVID-19 with acute respiratory failure (PaO2/FiO2 below 150).

Exclusion Criteria:

History of chronic cardiovascular, liver or/and kidney diseases. History of chronic pulmonary diseases with prolonged oxygen supplementation or domestic mechanical ventilation.

Pregnant women, Neoplastic diseases, Immunologic diseases Patients received immunomodulatory treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Xanthohumol reduces coronavirus-induced inflammatory response | one week after regular supplementation
  Xanthohumol possesses strong anti-inflammatory properties. It can reduce the production and secretion of pro-inflammatory cytokines. Additionally, it inhibits inflammatory-induced endothelial dysregulation and exerting antiangiogenic and anti-inflammatory effects.
Xanthohumol improves clinical course in critically ill COVID-19 patients | 28 days mortality
  Reduction the severity of inflammatory response should affect clinical course. Strong anti-inflammatory treatment can reduce a risk of poor outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Stepulak, Prof, Study Director — Rector of the Medical University of Lublin, Poland
Locations (1):
- Medical University of Lublin, Lublin, Poland